CLINICAL TRIAL: NCT03407209
Title: Compared Efficacy of Patient-controlled Epidural Analgesia With or Without Automatic Boluses
Acronym: FREE BOLI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-A01346-45
Record Dates: First submitted 2017-03-07; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Delivery
Keywords: Epidural analgesia; Patient Controlled Epidural Analgesia (PCEA); Patient Epidural Intermittent Bolus (PEIB); Local anesthetics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEIB - Use of local levobupivacaine anesthetics: 0.625 mg / ml (Sham Comparator): * automatic hourly bolus: 8ml (5mg) on 3 min
  * patient controlled bolus: 8ml (5mg) on 3 min
  * refractory period: 8min
  * continuous infusion: 0
  * maximum dose: 65mg/4h
  Interventions: Other: consumption of local anesthetic measurement
- FREE programming - levobupivacaine anesthetics: 0.625 mg / ml (Experimental): Epidural analgesia totally controlled by the patient
  * automatic hourly bolus: 0
  * patient controlled bolus: 8ml (5mg) on 3 min
  * refractory period: 8min
  * continuous infusion: 0
  * maximum dose: 65mg/4h
  Interventions: Other: consumption of local anesthetic measurement

INTERVENTIONS:
Other: consumption of local anesthetic measurement — consumption of local anesthetic measurement in both groups

SUMMARY:
Epidural analgesia is a significant feature of the everyday experience of the delivery room. Its benefits on the maternal experience and in terms of security has been widely demonstrated.

However, some women under epidural analgesia have experienced motor block, which has been found to contribute in the lengthening of the duration of labor, dystocia and instrumental delivery. Therefore, in recent years, reducing these side effects by modifying local anesthetics, concentration of local anesthetic and injected volume has been a priority, with one aim: optimize analgesia without motor blockage.

Although epidural analgesia was first provided by continuous epidural infusion, the efficacy of intermittent epidural bolus has been demonstrated. Small regularly spaced intermittent boluses lead to a more extensive and symmetrical spread of local anesthetic in the epidural space. These findings have led to a new kind of administration combining epidural intermittent boluses with patient-controlled boluses called PEIB (Patient Epidural Intermittent Bolus). On clinical grounds, PEIB is associated with reduced local anesthetic consumption and higher maternal satisfaction.

While PEIB is experimentally and clinically approved, incidence of maternal motor block and instrumental vaginal delivery don't decrease significantly with this programming. We hypothesized that automatic intermittent boluses can lead to an accumulation of local anesthetic overlapping with patient bolus. This accumulation can be the source of motor block, dystocia and instrumental delivery. Therefore, we propose to lead a monocentric prospective randomized study upon 308 patients in order to compare PEIB to epidural analgesia totally controlled by the patient. We expect a lower consumption of local anesthetic and a lower incidence of motor block, dystocia and instrumental delivery with the free automatic bolus programming.

DETAILED DESCRIPTION:
Local anesthetic used: levobupivacaine 0,625mg/ml

Solution prepared with 200 ml of levobupivacaine 0,625mg/ml associated with analgesic adjuvants: sufentanyl 50 micrograms and clonidine 75 micrograms.

Randomization between:

- PEIB:

* automatic hourly bolus: 8ml (5mg) on 3 min
* patient controlled bolus: 8ml (5mg) on 3 min
* refractory period: 8min
* continuous infusion: 0
* maximum dose: 65mg/4h

or

- FREE programming: epidural analgesia totally controlled by the patient

* automatic hourly bolus: 0
* patient controlled bolus: 8ml (5mg) on 3 min
* refractory period: 8min
* continuous infusion: 0
* maximum dose: 65mg/4h

Supervision and care consistent with french expert conference of the SFAR (Société Française d'Anesthésie-Réanimation) on management of women under epidural analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age >/= 18 years
* Nulliparous
* >35 weeks of amenorrhea
* In spontaneous or triggered labor

Exclusion Criteria:

* Contraindication for epidural analgesia (pre-partum hemostasis troubles, infection)
* Multiple pregnancy
* Fetal death in utero
* Programmed or in emergency caesarian

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women delivering
Enrollment: 462 (Actual)
Dates: Start 2016-11-06 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
consumption of local anesthetic | during delivery

SECONDARY OUTCOMES:
Incidence of motor block | during delivery
Incidence of dystocia | during delivery
Incidence of instrumental delivery | during delivery
Incidence of caesarian | during delivery
Incidence of oxytocin administration | during delivery
the evaluation of pain by a numerical scale rated from 0 to 10 | during delivery
Patient satisfaction with Likert type scale from A: excellent to E: catastrophic for the overall experience | during delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hopital, Caen, France

IPD SHARING:
Plan to Share IPD: No